CLINICAL TRIAL: NCT05176418
Title: IV Pulsed-Nicotine as a Model of Smoking: The Effects of Dose and Delivery Rate
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: HIC 2000032210
Record Dates: First submitted 2021-11-19; First posted 2022-01-04 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Intervention Model Description: This will be a double-blind, placebo-controlled study employing a mixed design: nicotine dose as the between-subject and delivery rate as the within-subject factors.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- delivery rate for nicotine dose 1mg/70kg (Active Comparator): delivery rate 50,35, 16.6 and 12.5 ug per second
  Interventions: Drug: low dose Nicotine
- Delivery rate for nicotine dose 0.2mg/70kg (Active Comparator): delivery rate 10,5, 3.3 and 2.5
  Interventions: Drug: high dose Nicotine

INTERVENTIONS:
Drug: low dose Nicotine — IV nicotine infused over different delivery rates
  Other Names: IV nicotine 1mg/70kg
  Arms: delivery rate for nicotine dose 1mg/70kg
Drug: high dose Nicotine — IV Nicotine infused over different delivery rates
  Other Names: IV Nicotine 0.2/70kg
  Arms: Delivery rate for nicotine dose 0.2mg/70kg

SUMMARY:
This project will examine the impact of the nicotine dose and delivery rate on nicotine's abuse potential, versus its potentially beneficial effects on smoking urges and withdrawal. Will use pulsed IV nicotine administration which closely matches nicotine delivery by inhaled tobacco use.

DETAILED DESCRIPTION:
Seventy smokers will be randomized to nicotine doses of either 0.2 or 1 mg per 70 kg body weight. Across 5 test sessions, within each dose group, participants will be randomly assigned to a sequence of 5 treatment conditions: placebo (saline) and 4 different delivery rates of nicotine. In each session, participants will receive either nicotine- or saline-pulsed infusions that will be delivered every 30 seconds for a total of 10 pulsed infusions. While receiving the pulsed infusions, participants will inhale a tobacco-flavored EC without nicotine, which will allow for a closer matching of the sensory aspects of inhaled tobacco use. There are four pulse duration conditions for the nicotine sessions: 2-, 4-, 6- and 8-second pulses. For those assigned to 1.0 mg/70kg nicotine dose, the pulse duration conditions correspond to nicotine delivery rates of 50, 25, 16.6, and 12.5 mcg nicotine/second. For those assigned to 0.2 mg/70 kg dose, the corresponding delivery rates will be 10, 5, 3.3 and 2.5 mcg nicotine/second. Participants in both nicotine dose groups will each have one placebo test session wherein they will receive 10 pulsed-saline infusions.

ELIGIBILITY:
Inclusion Criteria:

* Female and male, aged 21 to 55 years;
* past year daily cigarette use, verified by urine cotinine levels above 100 ng/ml -lifetime history of e-cigarette use; in good health as verified by medical history -screening examination, and screening laboratory tests
* women, -using acceptable birth control methods.

Exclusion Criteria:

* History of major medical or psychiatric disorders that the physician investigator deems as contraindicated for the participant to be in the study
* risk factors for EVALI (E-cigarette or Vaping Product Use-Associated Lung Injury) including history of lung diseases (e.g., asthma or COPD), vaping THC or CBD
* regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics)
* current alcohol or substance use disorder for any other recreational or prescription drugs other than nicotine
* for women, pregnant as determined by pregnancy screening, or breast feeding
* seeking (or undergoing) treatment for tobacco dependence or smoking; reported aversion to e-cigarettes, or tobacco flavored e-liquid.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Drug Effects Questionnaire mean score | up to five years
  The DEQ measures Good Drug Effect and consists of 11 questions with total score range from 0-100. Higher scores indicate more positive effects.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D.,Ph.D, Principal Investigator — Yale University
Locations (1):
- VA Healthcare System, West Haven, Connecticut, United States